CLINICAL TRIAL: NCT00293644
Title: A Randomized, Open-Label, Study of Pre-emptive Diclectin® Treatment for Severe Nausea and Vomiting of Pregnancy
Brief Title: Pre-emptive Treatment of Severe Nausea and Vomiting of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Duchesnay Inc. (Industry)
Responsible Party: Principal Investigator, Shinya Ito, Division Head, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000007791
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Hyperemesis Gravidarum; Pregnancy
Keywords: Pregnancy Complications; Hyperemesis Gravidarum; Diclectin; doxylamine succinate; pyridoxine hydrochloride
MeSH Terms: conditions — Hyperemesis Gravidarum; Pregnancy Complications | interventions — dicyclomine, doxylamine, pyridoxine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-emptive Treatment Group (Experimental): As soon as a patient becomes aware of the pregnancy, and before the Nausea and Vomiting of Pregnancy (NVP) starts, she will begin taking Diclectin®. When NVP starts, the dose will be adjusted to match symptoms.
  Interventions: Drug: Diclectin®
- Standard Treatment Group (Active Comparator): Women randomised to this arm will not receive any Diclectin® before symptoms appear, and will be advised to commence treatment only at first sign of nausea. The starting dose of Diclectin® will be 20mg (2 tablets) at bedtime.
  Interventions: Drug: Diclectin®
- Natural Course Group (No Intervention): A third group will be randomly matched from Motherisk NVP callers who did not participate in our pre-emptive intervention and experienced severe Nausea and Vomiting of Pregnancy/Hyperemesis Gravidarum (NVP/HG) in their previous pregnancy. This group will serve as a control group for the potential effect of the early counselling. (These women will have called for the first time after NVP symptoms (of any degree) started in the current pregnancy).

INTERVENTIONS:
Drug: Diclectin® — Participants will begin with an initial dose of 20mg (2 tablets), taken at bedtime. The dose of Diclectin® will be adjusted to match symptoms.
  Arms: Pre-emptive Treatment Group; Standard Treatment Group

SUMMARY:
The purpose of this study is to determine whether pre-emptive use of a delayed release combination of pyridoxine hydrochloride and doxylamine succinate (Diclectin®), before eruption of symptoms of Nausea and vomiting of pregnancy and hyperemesis gravidarum, will reduce the incidence of severe forms of this syndrome/HG.

DETAILED DESCRIPTION:
Nausea and vomiting of pregnancy (NVP) affects up to 80% of pregnant women, persists throughout pregnancy in 20% of women. 1%-3% of pregnant women experience the extreme form called hyperemesis gravidarum (HG), described as intractable vomiting associated with weight loss of more than 5% of pre-pregnancy weight, dehydration and electrolyte imbalances which may lead to hospitalization. Treatment involves administration of antiemetics once NVP occurs. Although there is wide evidence of fetal safety of several antiemetic medications, women and health professionals are often reluctant to use antiemetics due to a heightened misperception of teratogenic risk. Diclectin® is a prescription drug in Canada specifically indicated for treatment of NVP. Our preliminary research has shown Diclectin® to be effective for pre-emptive treatment for NVP symptoms in women who experienced severe NVP/HG in their previous pregnancy. This study will evaluate the effectiveness of Diclectin as a pre-emptive treatment for NVP and HG in a randomized controlled trial. In the Pre-emptive Treatment Group, as soon as a patient becomes aware of the present pregnancy, and before the NVP starts, she will take an initial Diclectin® dose, followed by standard dosing to match symptoms once NVP develops. In the Standard Treatment Group women will take Diclectin® only at appearance of symptoms. A natural history control group will also be included. This study will determine whether pre-emptive use of Diclectin will reduce the incidence of severe forms of this syndrome/HG.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy of less than 9 weeks gestation with no symptoms of NVP
* Not pregnant
* Include all women with severe NVP/HG in a previous pregnancy regardless of outcome
* Severe NVP/HG in a previous pregnancy verbally confirmed by the initial recruitment intake questionnaire or previous pregnancy history of NVP/HG section (duration, severity, treatments, and hospitalisation)
* Verbally agree to participate in the study and send back rhe informed consent form
* Sufficient French or English language skills to understand the questionnaire and assessment material
* Women who agree to take Diclectin®
* Women can enrol with a consecutive pregnancy, if the study is still ongoing

Exclusion Criteria:

* Women who refuse to participate in the study or to send back the signed consent form
* Women with insufficient French or English language skills to understand the questionnaire and assessment material
* Women their first pregnancy and those who havn't suffered severe NVP/HG in previous pregnancy
* Gestational age beyond 9w+0d weeks of pregnancy
* Pregnant women who already suffer symptoms of NVP
* Pregnant women with known hypersensitivities to Diclectin®
* Women who do not agree to take Diclectin®
* Women who suffer symptoms of pyelonephritis, thyrotoxicosis, gestational trophoblastic neoplasia
* Pregnant women less than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-02; Primary Completion 2012-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of severe NVP (defined by PUQE score >12), or HG (defined by PUQE score >12 plus hospitalization), as compared among the 3 groups. | Follow-up in all groups will be continued monthly until delivery. An additional follow-up telephone interview will be done at approximately 6 months post delivery.

SECONDARY OUTCOMES:
Comparing the incidence of NVP/HG in present pregnancy with incidence of NVP/HG from the previous pregnancies. | Follow-up in all groups will be continued monthly until delivery. An additional follow-up telephone interview will be done at approximately 6 months post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Shinya Ito, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Preemptive treatment of nausea and vomiting of pregnancy: results of a randomized controlled trial. — http://www.ncbi.nlm.nih.gov/pubmed/23476657